CLINICAL TRIAL: NCT00053209
Title: Phase II Trial Of Pemetrexed Disodium And Gemcitabine In Advanced Urothelial Cancer
Brief Title: Pemetrexed Disodium and Gemcitabine in Treating Patients With Advanced Cancer of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269302; ECOG-E4802
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; transitional cell carcinoma of the bladder; recurrent bladder cancer; stage III bladder cancer; stage IV bladder cancer; anterior urethral cancer; posterior urethral cancer; recurrent urethral cancer; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed Disodium and Gemcitabine (Experimental): Pemetrexed disodium 500 mg/m2 followed by gemcitabine 1000 mg/m2 on day 1 and gemcitabine 1000 mg/m2 on day 8 of a 21-day cycle for a maximum of 6 cycles
  Interventions: Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Pemetrexed disodium may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining pemetrexed disodium with gemcitabine may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining pemetrexed disodium with gemcitabine in treating patients who have advanced cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with previously untreated advanced cancer of the urothelium treated with pemetrexed disodium and gemcitabine.
* Determine the toxicity of this regimen in these patients.

Secondary

* Determine the overall survival and time to progression in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive pemetrexed disodium IV over 10 minutes on day 1 and gemcitabine IV over 30 minutes on days 1 and 8. Patients also receive cyanocobalamin intramuscularly once every 9 weeks and folic acid orally once daily beginning on day -6 and continuing until 3 weeks after the completion of study therapy. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 24-46 patients will be accrued for this study within 15 -18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer of the urothelium (renal pelvis, ureter, bladder, or urethra)

  * Any of the following types:

    * Transitional cell carcinoma (TCC)
    * Mixed histologies containing a component of TCC
    * Non-TCC of the urothelium (renal pelvis, ureter, bladder, or urethra)
* Progressing regional or metastatic disease
* Measurable disease
* No clinical evidence of CNS metastases
* No evidence of clinically significant (by physical exam or plain film) third-space fluid collections (pleural effusions or ascites)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic

* AST no greater than 3 times upper limit of normal (ULN)
* Bilirubin no greater than 1.5 times ULN

Renal

* Creatinine clearance at least 45 mL/min

Cardiovascular

* No history of severe cardiovascular disease (i.e., American Heart Association class III or IV heart disease)
* No uncontrolled congestive heart failure
* No ventricular dysrhythmias

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active unresolved infection
* No other prior malignancy unless curatively treated and disease free for an appropriate (disease-specific) period of time
* Able and willing to receive folic acid and cyanocobalamin supplementation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior systemic biologic response modifier therapy

Chemotherapy

* No prior systemic chemotherapy for metastatic disease
* More than 1 year since prior neoadjuvant or adjuvant chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No prior pelvic radiotherapy
* No concurrent radiotherapy

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* More than 7 days since prior parenteral antibiotics
* No salicylates for 2 days before, during, and for 2 days after administration of pemetrexed disodium
* No nonsteroidal anti-inflammatory drugs for at least 5 days before, during, and for 2 days after administration of pemetrexed disodium

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-08-10 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Response as measured by RECIST criteria | Assessed every 6 weeks

SECONDARY OUTCOMES:
Time to disease progression | Assessed every 6 weeks
Overall survival | Assessed every 3 months for 2 years, then every 6 months for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreicer, MD, FACP, Study Chair — The Cleveland Clinic
Locations (121):
- United States (121):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Watson Clinic, LLC, Lakeland, Florida
  - Hematology and Oncology of Northeast Georgia, Athens, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Saint Joseph Regional Medical Center - Plymouth Campus, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Union Hospital Cancer Center at Union Hospital, Elkton, Maryland
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Hospital, Woodbury, Minnesota
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Mountainside Hospital Cancer Center, Montclair, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, P. C., Lemoyne, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Cancer Care Institute of Carolina at Aiken Regional Medical Centers, Aiken, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Erlanger Cancer Center, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Cancer Care Center at Holy Family Memorial Medical Center, Manitowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Dreicer R, Li H, Cooney MM, Wilding G, Roth BJ; Eastern Cooperative Oncology Group. Phase 2 trial of pemetrexed disodium and gemcitabine in advanced urothelial cancer (E4802): a trial of the Eastern Cooperative Oncology Group. Cancer. 2008 Jun 15;112(12):2671-5. doi: 10.1002/cncr.23503. PMID 18459175
- [Result] Li S, Dreicer R, Roth B, et al.: Phase II trial of pemetrexed disodium and gemcitabine in advanced carcinoma of the urothelium (E4802): a trial of the Eastern Cooperative Oncology Group. [Abstract] J Clin Oncol 25 (Suppl 18): A-5079, 254s, 2007.